CLINICAL TRIAL: NCT03882892
Title: Long-Term, Safety and Tolerability Study of SCH 58235 or Placebo in Addition to Atorvastatin in Subjects With Primary Hypercholesterolemia
Brief Title: Long-Term Safety and Tolerability of Ezetimibe (SCH 58235, MK-0653) With Atovastatin (P02154, MK-0653-017)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P02154; MK-0653-017 (Other: Merck Protocol Number); P02154 (Other: Schering-Plough Protocol Number)
Record Dates: First submitted 2019-03-19; First posted 2019-03-20 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo + Atorvastatin (Placebo Comparator): Participants who received placebo in the parent study (P00692) receive placebo (blinded) + atorvastatin (10 mg/day; open-label) in this study.
  Interventions: Drug: Atovastatin; Drug: Placebo
- Ezetimibe + Atorvastatin (Experimental): Participants who received ezetimibe + atorvastatin, or atorvastatin alone, in the parent study (P00692) receive ezetimibe (blinded) + atorvastatin (10 mg/day; open-label) in this study.
  Interventions: Drug: Ezetimibe; Drug: Atovastatin

INTERVENTIONS:
Drug: Ezetimibe — Ezetimibe 10 mg tablets
  Other Names: SCH 58235
  Arms: Ezetimibe + Atorvastatin
Drug: Atovastatin — Atorvastatin 10, 20, and 40 mg tablets at a daily dose of 10 to 80 mg
Drug: Placebo — Placebo tablets matched to ezetimibe
  Arms: Placebo + Atorvastatin

SUMMARY:
The purpose of this study is to examine the long-term safety and tolerability of ezetimibe (SCH 58235) 10 mg once daily or placebo in combination with atorvastatin (10 to 80 mg/day) for up to 12 consecutive months in participants with primary hypercholesterolemia.

DETAILED DESCRIPTION:
This study is a long-term extension study of the protocol P00692 parent study.

ELIGIBILITY:
Inclusion Criteria:

* Has successfully completed the 12-week double-blind, efficacy and safety parent study (P00692).
* If female, has a negative pregnancy test prior to study entry and, if of childbearing potential, agrees to practice an effective barrier method of birth control for the duration of the study and for 30 days after the last statin dose.
* If postmenopausal female receiving hormone therapy, a stable estrogen (ERT), estrogen/progestin (HRT) or raloxifene regimen must be maintained during the study period.
* Is willing to continue to follow their prescribed National Cholesterol Education Program (NCEP) Step 1 diet for the duration of the study.

Exclusion Criteria:

* Has discontinued from the parent study (P00692) prior to study completion.
* Is in a situation, or has any condition which, in the opinion of the investigator may interfere with optimal participation.
* Is a pregnant or lactating female.
* Is human immunodeficiency virus (HIV) positive.

Ages: 18 Years to 86 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2001-02-02 (Actual); Primary Completion 2002-08-08 (Actual); Study Completion 2002-08-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Experiencing ≥1 Adverse Event (AE) | Up to 12 months
Percentage of Participants Discontinuing from Study Treatment due to an Adverse Event (AE) | Up to 12 months

SECONDARY OUTCOMES:
Mean Percent Change from Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline and 1.5, 3, 6, 9, and 12 months
Mean Percent Change from Baseline in High-Density Lipoprotein Cholesterol (HDL-C) | Baseline and 1.5, 3, 6, 9, and 12 months
Mean Percent Change from Baseline in Triglyceride Levels | Baseline and 1.5, 3, 6, 9, and 12 months
Mean Percent Change from Baseline in Total Cholesterol (TC) | Baseline and 1.5, 3, 6, 9, and 12 months
Mean Percent Change from Baseline in Calculated Low-Density Lipoprotein Cholesterol (LDL-C) | Baseline and 1.5, 3, 6, 9, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ballantyne CM, Lipka LJ, Sager PT, Strony J, Alizadeh J, Suresh R, Veltri EP. Long-term safety and tolerability profile of ezetimibe and atorvastatin coadministration therapy in patients with primary hypercholesterolaemia. Int J Clin Pract. 2004 Jul;58(7):653-8. doi: 10.1111/j.1368-5031.2004.00278.x. PMID 15311720